CLINICAL TRIAL: NCT00056953
Title: Peer Mentors for Early Adolescents in HIV-Affected Families
Brief Title: Peer Mentors for Adolescents in HIV Affected Families
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01HD37350-3; 5R01HD037350 (NIH)
Record Dates: First submitted 2003-03-26; First posted 2003-03-27 (Estimated); Last update posted 2005-07-29 (Estimated); Status verified 2005-07

CONDITIONS: Adolescent Behavior; Health Behavior; HIV Seronegativity
Keywords: health behavior; adolescent behavior; peer mentoring
MeSH Terms: conditions — Adolescent Behavior; Health Behavior

INTERVENTIONS:
Behavioral: Peer mentoring program

SUMMARY:
This study will evaluate the effectiveness of a peer mentoring program designed for youths ages 9 to 15 whose parents or guardians are HIV infected. The program will focus on the youths' mental health, school performance, alcohol and drug use, personal and social behaviors, and behaviors that might expose them to HIV. The study is expected to enroll predominantly minority youth.

DETAILED DESCRIPTION:
This study will conduct an efficacy trial of peer mentoring for a high-risk, predominantly minority population of 9- to 15-year-old youths whose parents are HIV infected. The study will also determine mechanisms (mediating variables) through which peer mentoring improves outcomes for the mentees, for example, consistency and continuity of relationship, teaching/role modeling, emotional support/empathy, advocacy, and behavioral reinforcement. After the conclusion of the efficacy trial, the study will continue through naturalistic longitudinal research for an additional 2 years in order to examine the long-term outcomes of peer mentoring.

Participants are randomized to either the peer mentoring program or a control condition (a recreation program). Surveys are conducted at entry into the study, at 6 months, 1 year, and then annually for 2 years. Youths will also participate in focus groups. The surveys and focus groups will assess the youths' psychological functioning, academic adjustment, alcohol and drug use, HIV risk behaviors, delinquent/violent behaviors, peer relationships, prosocial activities, and coping/problem-solving skills. The study will also evaluate family outcomes, including parent/guardian functioning and improved permanency planning.

ELIGIBILITY:
Inclusion Criteria

* HIV infected parent or guardian
* No previous involvement in the mentoring program
* Adolescent assent
* Parental consent

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160
Dates: Start 1999-09; Study Completion 2004-11

PRIMARY OUTCOMES:
substance use; association with substance using peers

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Magura, Ph.D., Principal Investigator — National Development and Research Institutes, Inc.
Locations (1):
- Health People, New York, New York, United States

REFERENCES:
- [Result] Rosenblum A, Magura S, Fong C, Cleland C, Norwood C, Casella D, Truell J, Curry P. Substance use among young adolescents in HIV-affected families: resiliency, peer deviance, and family functioning. Subst Use Misuse. 2005;40(5):581-603. doi: 10.1081/ja-200030816. PMID 15887592